CLINICAL TRIAL: NCT02815657
Title: A Single Randomized, Open,Cross-over, Phase I Study to Access the Drug-drug Interaction of SP2086 and Valsartan
Brief Title: The Drug-drug Interaction of SP2086 and Valsartan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR-SP-106
Record Dates: First submitted 2016-01-03; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes
Keywords: SP2086; Valsartan; Drug-drug Interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SP2086 and Valsartan (Active Comparator): All subject were randomized into two groups,and the drugs will be administered according to the AB and BA sequences,all subjects must completed the two stages(A and B).The A sequence was that Valsartan was taken at 160mg qd on Days1-Day12; SP2086 will be administered orally (by mouth) as 200mg on Days 8-Day12.The B sequence was that SP2086 was taken at 200mg qd dose on Days 8-Day12.There were 6 days washout period between the two stages.The whole study needs 31 days.This group patient was given treatment from A stage to B stage.
  Interventions: Drug: SP2086; Drug: Valsartan
- Valsartan and SP2086 (Active Comparator): All subject were randomized into two groups,and the drugs will be administered according to the AB and BA sequences,all subjects must completed the two stages(A and B).The A sequence was that Valsartan was taken at 160mg qd on Days1-Day12; SP2086 will be administered orally (by mouth) as 200mg on Days 8-Day12.The B sequence was that SP2086 was taken at 200mg qd dose on Days 8-Day12.There were 6 days washout period between the two stages.The whole study needs 31 days.This group patient was given treatment from B stage to A stage.
  Interventions: Drug: SP2086; Drug: Valsartan

INTERVENTIONS:
Drug: SP2086 — The A sequence was that Valsartan was taken at 160mg qd on Days1-Day12; SP2086 will be administered orally (by mouth) as 200mg on Days 8-Day12.The B sequence was that SP2086 was taken at 200mg qd dose on Days 8-Day12
Drug: Valsartan — The A sequence was that Valsartan was taken at 160mg qd on Days1-Day12; SP2086 will be administered orally (by mouth) as 200mg on Days 8-Day12.The B sequence was that SP2086 was taken at 200mg qd dose on Days 8-Day12

SUMMARY:
The purpose of the study is to investigate the potential interaction between SP2086 and Valsartan after multiple oral doses treatment in healthy adult volunteers.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned) single-center and cross-over study of SP2086 and Valsartan in healthy adult volunteers. All subject were randomized into two groups, and the drugs will be administered according to the AB and BA sequences, all subjects must completed the two stages(A and B). The A sequence was that Valsartan was taken at 160mg qd on Days1-Day12; SP2086 will be administered orally (by mouth) as 200mg on Days 8-Day12.The B sequence was that SP2086 was taken at 200mg qd dose on Days 8-Day12.There were 6 days washout period between the two stages. The whole study needs 31 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index(BMI) between 19 and 24 Kg/m2
* Had signed the informed consent himself or herself.

Exclusion Criteria:

* Have the abnormal lab or other examination results and the change have clinical significance.
* History of or current clinically significant medical illness as determined by the Investigator.
* Have a family history of thyroid cancer, submandibular gland cancer or long QT syndrome
* Known allergy to SP2086 or Glyburide or any of the excipients of the formulation of SP2086 or Glyburide.
* History of using the sulfa or sulfonylureas or DPP-IVor GLP-1 drugs or other similar structure drugs.
* History of severe unconsciousness hypoglycemia
* History of any surgery prior to screening in 6 months.
* History of blood donation≥400 mL prior to screening in 3 months or participate in blood donation,or by blood transfusion in one month.
* History of participate any drug or medical device prior to screening in 3 months.
* Within a month before the screening using any prescription drugs, over-the-counter drugs, Chinese herbal medicine (especially oral antidiabetics drugs) or food supplements( vitamins).
* 2 days before the randomization ,the patients can not ban alcohol, tobacco, or reference food or drink containing caffeine or xanthine , or vigorous exercise, or there are other factors that can affect drug absorption, distribution, metabolism and excretion.
* The hepatitis B surface antigen, hepatitis c antibody, HIV antibody and syphilis antibody was positive.
* Pregnancy or lactation women, or a fertility male or female is not willing to contraception during test.
* Researchers considered that there was any situation that may cause the participants can't finish this study or bring any obvious risk to subjects.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to Day 31
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The maximum plasma concentration (Cmax) of SP2086 acid | up to Day 31
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The maximum plasma concentration (Cmax) of valsartan | up to Day 31
  Cmax (a measure of the body's exposure to valsartan) will be compared before and after administration of multiple doses of valsartan
The area under the plasma concentration-time curve (AUC) of SP2086 | up to Day 31
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of SP2086 acid | up to Day 31
  AUC (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of valsartan | up to Day 31
  AUC (a measure of the body's exposure to valsartan) will be compared before and after administration of multiple doses of valsartan

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 31

CONTACTS AND LOCATIONS:
Overall Officials: XiaoLan Yong, P.H.D, Principal Investigator — People's Liberation Army General Hospital of Chengdu Military Region
Locations (1):
- People's Liberation Army General Hospital of Chengdu Military Region, Chengdu, China